CLINICAL TRIAL: NCT04782791
Title: A Prospective, Randomized, Controlled Phase II Evaluation of Nivolumab, S-1 Combined With Oxaliplatin (Nivo+SOX) Versus Nivolumab (Nivo) as Neoadjuvant Therapy in Patients With Locally Advanced Gastric Adenocarcinoma (RESONANCE-Ⅲ Study)
Brief Title: Nivolumab, S-1 Combined With Oxaliplatin Versus Nivolumab as Neoadjuvant Therapy in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3
Record Dates: First submitted 2021-01-25; First posted 2021-03-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer; Chemotherapy Effect
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivo + SOX (Experimental): Nivolumab plus SOX
  Interventions: Drug: Nivolumab plus SOX; Procedure: Gastrectomy
- Nivo (Active Comparator): Nivolumab
  Interventions: Drug: Nivolumab; Procedure: Gastrectomy

INTERVENTIONS:
Drug: Nivolumab plus SOX — The preoperative therapy consists of three-week cycles of intravenously administered nivolumab 360mg and oxaliplatin 130mg/m2 on day 1, and orally administered S-1 40-60 mg twice a day (BID) on day 1 to 14. The dose of S-1 depends on body surface area (BSA): BSA<1.25 m2, 40mg; 1.25<BSA<1.50 m2, 50mg; BSA>1.50 m2, 60mg. Day 15 to day 21 is the rest period.
  Other Names: Nivo + SOX
  Arms: Nivo + SOX
Drug: Nivolumab — The preoperative therapy consists of three-week cycles of intravenously administered nivolumab 360mg on day 1.
  Other Names: Nivo
  Arms: Nivo
Procedure: Gastrectomy — A standard D2 radical laparoscopic gastrectomy according to the CSCO clinical guidelines for the diagnosis and treatment of gastric cancer is planned 3-4 weeks after the last cycle of preoperative therapy.

SUMMARY:
The trial is a prospective, randomized, controlled phase Ⅱ study which will be conducted in Chinese PLA General Hospital, Beijing, China. Patients with eligibility will enrolled and assigned into either group A for 9 weeks of nivolumab, S-1 combined with oxaliplatin (Nivo+SOX) followed by D2 surgery and group B for 9 weeks of nivolumab followed by D2 surgery. The primary endpoint is the safety assessed by recording adverse events and the secondary endpoints are response rate, disease control rate, pathological complete response rate, D2 rate and R0 rate.

ELIGIBILITY:
Inclusion Criteria:

* Non-bedridden, aged 18 to 70 years old;
* Eastern Cooperative Oncology Group (ECOG) score is 0 to 1;
* Histologically confirmed gastric adenocarcinoma;
* Have evaluable lesions based on RECIST 1.1;
* Stage III (cT3-4aN1-3 M0, American Joint Committee on Cancer (AJCC) TNM staging system 8th edition) gastric cancer confirmed by enhanced computer tomography (enhanced CT) and laparoscopic exploration (endoscopic ultrasonography (EUS) and magnetic resonance imaging (MRI) if necessary);
* The surgeon have the ability to complete standard D2 radical gastrectomy and the gastrectomy can be tolerated by the patient;
* Laboratory test criteria: peripheral blood hemoglobin (Hb) ≥ 90 g/L, neutrophil absolute count ≥ 3× 109 /L, platelet count (PLT) ≥ 100× 109 /L, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN), total bilirubin ≤ 1.5×ULN, serum creatinine (SCr) ≤ 1.5×ULN, and serum albumin (ALB) ≥ 30 g/L;
* Patients with heart disease, echocardiogram showing that the left ventricular ejection fraction ≥ 50%, electrocardiogram (ECG) is basically normal within 4 weeks before operation and with no obvious symptoms are acceptable;
* There is no serious underlying disease that could lead to an expected life expectancy < 5 years;
* Willing to sign the informed consent for participation and publication of results.

Exclusion Criteria:

* Human epidermal growth factor receptor 2 (HER2)-positive or indeterminate G/GEJ cancer;
* Pregnant or lactating women;
* Positive pregnancy test for women in childbearing age. Menopausal women without menstruation for at least 12 months can be regarded as women with no possibility of getting pregnant;
* Refusal of birth control during the study;
* Prior chemotherapy, radiotherapy or immunotherapy;
* History of other malignant diseases in the last 5 years (except for cervical carcinoma in situ);
* History of uncontrolled central nervous system diseases, which could influence the compliance;
* History of severe liver diseases (Child-Pugh class C), renal diseases (endogenous creatinine clearance rate (Ccr) ≤ 50 ml/min or SCr > 1.5 ULN) or respiratory diseases; Uncontrolled diabetes and hypertension; Clinically severe heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure, uncontrolled arrhythmia requiring drug intervention, or a history of myocardial infarction in the last 6 months;
* History of dysphagia, complete or partial gastrointestinal obstruction, active gastrointestinal bleeding and gastrointestinal perforation;
* On steroid treatment after organ transplant;
* With uncontrolled severe infections;
* Known dihydropyrimidine dehydrogenase deficiency (DPD);
* Anaphylaxis to any research drug ingredient;
* Known peripheral neuropathy (> NCI-CTC AE 1). Patients with only disappearance of deep tendon reflex need not to be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 years
  The safety is assessed by recording adverse events.

SECONDARY OUTCOMES:
RR | 2 years
  Response rate, defined as the rate of patients who achieve CR or PR according to the RESIST 1.1.
DCR | 2 years
  Disease control rate, defined as the rate of patients who achieve CR, PR or PD according to the RESIST 1.1.
pCR rate | 2 years
  Pathological complete response rate, defined as the rate of patients achieving pathological complete response.
D2 rate | 2 years
  The rate of patients who received D2 radical gastrectomy.
R0 rate | 2 years
  The rate of patients who received R0 resection.